CLINICAL TRIAL: NCT03294538
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Design, Multiple-Site Study to Evaluate the Therapeutic Equivalence of Estradiol Vaginal Cream USP, 0.01% (Teva Pharmaceuticals, USA) to Estrace® Estradiol Vaginal Cream, USP, 0.01% (Warner Chilcott) in the Treatment of Atrophic Vaginitis
Brief Title: Study to Evaluate Equivalence of Estradiol Vaginal Cream 0.01% to Estrace® Cream 0.01% in Atrophic Vaginitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 71436001
Record Dates: First submitted 2017-09-20; First posted 2017-09-27 (Actual); Results first posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Atrophic Vaginitis
MeSH Terms: conditions — Atrophic Vaginitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Generic Estradiol Vaginal Cream USP, 0.01% (Experimental): Participants were to self-administer 2 grams (g) of generic Estradiol Vaginal Cream USP, 0.01% once daily at approximately the same time of the day for 7 consecutive days.
  Interventions: Drug: Generic Estradiol Vaginal Cream USP, 0.01%
- Estrace Vaginal Cream USP, 0.01% (Active Comparator): Participants were to self-administer 2 g of Estrace Vaginal Cream USP, 0.01% once daily at approximately the same time of the day for 7 consecutive days.
  Interventions: Drug: Estrace® Vaginal Cream USP, 0.01%
- Vehicle Vaginal Cream (Placebo Comparator): Participants were to self-administer 2 g of vehicle vaginal cream once daily at approximately the same time of the day for 7 consecutive days.
  Interventions: Drug: Vehicle Vaginal Cream

INTERVENTIONS:
Drug: Generic Estradiol Vaginal Cream USP, 0.01% — Vaginal cream, generic formulation of the brand product.
  Arms: Generic Estradiol Vaginal Cream USP, 0.01%
Drug: Estrace® Vaginal Cream USP, 0.01% — Vaginal cream, brand product.
  Arms: Estrace Vaginal Cream USP, 0.01%
Drug: Vehicle Vaginal Cream — Vaginal cream, placebo. Has no active ingredient
  Arms: Vehicle Vaginal Cream

SUMMARY:
The objectives of this study were to evaluate the therapeutic equivalence of the Test formulation, generic Estradiol Vaginal Cream United States Pharmacopoeia (USP), 0.01% (Teva Pharmaceuticals, United States of America) to the marketed product, Estrace® Cream estradiol vaginal cream USP, 0.01% (Warner Chilcott) in participants with atrophic vaginitis; to demonstrate the superiority of the Test and Reference (active) treatments over Placebo (vehicle) cream in participants with atrophic vaginitis; and to compare the safety of Test, Reference, and Placebo treatments in participants with atrophic vaginitis.

DETAILED DESCRIPTION:
Systemic (oral or transdermal patch administration) estrogen therapies have been shown to effectively treat symptoms of atrophic vaginitis but bear undesirable side effects including increased risk of heart attacks, stroke, endometrial cancer, and breast cancer. Topical therapies (creams and transvaginal delivery systems) provide low doses of estrogen to the vaginal mucosa to provide local relief for the symptoms of atrophic vaginitis, while reducing the unwanted side effects associated with systemic delivery systems. Low dose, topical estrogen therapy is considered most appropriate and convenient for the treatment of vaginal symptoms associated with menopause, particularly when other symptoms including bone loss or vasomotor dysfunction do not need to be targeted.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form (ICF) that meets all criteria of current Food and Drug Administration (FDA) regulations.
* Females aged 30-75 years inclusive who are postmenopausal, defined as follows:
* At least 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum follicle-stimulating hormone (FSH) level of >40 milli-international units per milliliter (mIU/mL); at least 6 weeks post-surgical bilateral oophorectomy, with or without hysterectomy; or hysterectomy without oophorectomy if of age that the Investigator believes would have been naturally reached 12 months of spontaneous amenorrhea.
* Vaginal pH >5.0.
* At least 1 of the following participant self-assessed moderate to severe symptoms of vulvar and vaginal atrophy (VVA) from the following list that is identified by the participant as being most bothersome to her:

  1. Vaginal Dryness
  2. Vaginal and/or vulvar irritation/itching
  3. Dysuria
  4. Vaginal pain or bleeding associated with sexual activity, provided that participant is currently sexually active and plans to remain so throughout study.
* "Normal" Screening mammogram completed within 9 months prior to Screening in all participants >40 years old.
* Normal clinical breast examination at the Screening Visit.
* Documented papanicolaou (PAP) smear conducted within the previous 12 months with no findings that the Investigator believes would contraindicate the use of topical vaginal estradiol.
* Participants with an intact uterus should have vaginal ultrasonography results to confirm an inactive endometrial lining, defined as endometrial thickness less than 4 millimeters (mm).

Exclusion Criteria:

1. Females younger than 30 years of age or older than 75 years of age.
2. Participants with a Serum follicle-stimulating hormone (FSH) level of ≤40 mIU/mL at Screening.
3. Greater than 5% superficial cells on vaginal cytology.
4. Vaginal pH ≤5.
5. Significant history or current evidence of chronic infectious disease, system disorder, organ disorder (including significant liver/kidney impairment) or other medical condition that in the Investigator's opinion would place the study participant at undue risk by participation or could jeopardize the integrity of the study evaluations.
6. Participants with an intact uterus should have vaginal ultrasonography results to confirm an inactive endometrial lining. Participants with an endometrial thickness equal to or greater than 4 mm.
7. Documented PAP smear conducted within the previous 12 months with findings that the Investigator believes would contraindicate the use of topical vaginal estradiol.
8. Participants with known concurrent vaginal infections including but not limited to:

   Candida albicans, Trichomonas vaginalis, Chlamydia trachomatis, Neisseria gonorrhea, or Gardnerella vaginalis.
9. Participants with active vaginal herpes simplex infection or have had an outbreak within 30 days of the first dosing day.
10. Participants with known, suspected, or current history of carcinoma of the breast. All participants over the age of 40 must have had a mammogram performed within 9 months of the study start and all participants will have a physical breast exam performed at Screening.
11. Participants with known, suspected or current history of hormone dependent tumor.
12. Participants with baseline systolic blood pressure of >150 millimetres of mercury (mmHg) and/or diastolic pressure >90 mmHg.
13. Any participant with undiagnosed vaginal bleeding or significant risk factors for endometrial cancer.
14. Any history of estrogen-dependent neoplasia (for example, endometrial cancer).
15. History of acute thrombophlebitis or thromboembolic disorder.
16. Any current or recent (within the previous 6 months) genital bleeding of unknown etiology.
17. Any prescription treatment or over-the-counter (OTC) or natural remedies for vaginal dryness/irritation within 28 days of Screening. Products used for lubrication during sexual intercourse within 7 days of Screening.
18. Participants whose fasting triglyceride levels are greater than 350 mg/dL.
19. Any participant with a history of radiation therapy or recent (within previous 6 weeks) surgical therapy to the vaginal or cervical areas.
20. Any known or suspected allergies that in the Investigator's opinion would compromise the safety of the participant.
21. Participants who have used vaginal hormonal products (rings, creams, gels) within the 28 days prior to Screening.
22. Any participant who has used transdermal estrogen and/or progestin therapy within the 28 days prior to Screening.
23. Participants who have used oral estrogen and/ or progestin therapy or intrauterine progestin therapy within the 56 days prior to Screening.
24. Participants who have used progestin implants or estrogen alone injectable drug therapy within the 3 months before Screening.
25. Participants who have used estrogen pellet therapy or progestin injectable drug therapy within the 6 months before Screening.
26. Participants who, in the opinion of the Investigator, would be non-compliant with the requirements of the study protocol.
27. Participants who are unable or unwilling to give informed consent.
28. Receipt of any drug as part of a research study within 30 days prior to Screening.
29. Participants who have participated in this study previously.

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 663 (Actual)
Dates: Start 2016-05-18 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Teva Pharmaceuticals USA
Locations (44):
- United States (44):
  - Site Number 44, Tucson, Arizona
  - Site Number 17, Tucson, Arizona
  - Site Number 31, La Mesa, California
  - Site Number 11, Sacramento, California
  - Site Number 05, San Diego, California
  - Site Number 15, San Diego, California
  - Site Number 25, Colorado Springs, Colorado
  - Site Number 01, Denver, Colorado
  - Site Number 14, Denver, Colorado
  - Site Number 18, New London, Connecticut
  - Site Number 06, Jupiter, Florida
  - Site Number 13, Lake Worth, Florida
  - Site Number 27, Miami, Florida
  - Site Number 40, Miami, Florida
  - Site Number 20, Miami, Florida
  - Site Number 39, Miami, Florida
  - Site Number 38, Miami, Florida
  - Site Number 30, Miami Lakes, Florida
  - Site Number 08, New Port Richey, Florida
  - Site Number 03, Ormond Beach, Florida
  - Site Number 45, Port Saint Lucie, Florida
  - Site Number 10, Sarasota, Florida
  - Site Number 19, St. Petersburg, Florida
  - Site Number 02, West Palm Beach, Florida
  - Site Number 29, Roswell, Georgia
  - Site Number 22, Savannah, Georgia
  - Site Number 21, Wichita, Kansas
  - Site Number 33, Metairie, Louisiana
  - Site Number 16, Kalamazoo, Michigan
  - Site Number 34, Saginaw, Michigan
  - Site Number 35, Lincoln, Nebraska
  - Site Number 12, Lawrenceville, New Jersey
  - Site Number 26, Plainsboro, New Jersey
  - Site Number 36, Raleigh, North Carolina
  - Site Number 04, Winston-Salem, North Carolina
  - Site Number 37, Winston-Salem, North Carolina
  - Site Number 07, Columbus, Ohio
  - Site Number 24, Englewood, Ohio
  - Site Number 28, West Chester, Ohio
  - Site Number 23, Bluffton, South Carolina
  - Site Number 41, Mt. Pleasant, South Carolina
  - Site Number 43, Myrtle Beach, South Carolina
  - Site Number 32, Dallas, Texas
  - Site Number 09, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The populations for this study included the Safety Population, the modified Intent-to-Treat (mITT) population, and the Per-Protocol (PP) Population.
Pre-assignment Details: Following the 14-day screening period, participants who continued to meet the inclusion/exclusion (I/E) criteria were randomly assigned to treatment on a 2:2:1 ratio of generic Estradiol Vaginal Cream United States Pharmacopoeia (USP), 0.01%; Estrace Vaginal Cream USP, 0.01%; or vehicle vaginal cream.
Groups:
- Generic Estradiol Vaginal Cream USP, 0.01%: Participants were to self-administer 2 g of generic Estradiol Vaginal Cream USP, 0.01% once daily at approximately the same time of the day for 7 consecutive days.
Period: Overall Study
Arm/Group | Generic Estradiol Vaginal Cream USP, 0.01% | Estrace Vaginal Cream USP, 0.01% | Vehicle Vaginal Cream
Started | 268 | 262 | 133
Safety Population (All participants who were randomized and administered at least 1 dose of study drug) | 267 | 262 | 132
mITT Population (mITT population, administered at least 1 dose of study drug, and had a post-randomization evaluation) | 267 | 262 | 132
PP Population (Met I/E criteria, didn't develop concurrent vaginal infection, completed Day 8 visit, took 6-8 doses) | 244 | 227 | 126
Completed | 263 | 257 | 131
Not Completed | 5 | 5 | 2
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Outside of Visit Window | 4 | 4 | 1

BASELINE CHARACTERISTICS:
Population: All participants who were randomized and administered at least 1 dose of study drug (Safety Population).
Groups:
- Total: Total of all reporting groups
Arm/Group | Generic Estradiol Vaginal Cream USP, 0.01% | Estrace Vaginal Cream USP, 0.01% | Vehicle Vaginal Cream | Total
Number analyzed (Participants) | 267 | 262 | 132 | 661
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.5 (6.4) | 59.5 (6.5) | 60.8 (5.6) | 59.9 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 267 | 262 | 132 | 661
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 79 | 88 | 42 | 209
  Not Hispanic or Latino | 188 | 174 | 90 | 452
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 0 | 3
  Asian | 5 | 3 | 0 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 25 | 24 | 10 | 59
  White | 235 | 232 | 121 | 588
  More than one race | 0 | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Percent of Basal/Parabasal Cells [Mean (Standard Deviation); unit: percent of cells] — Population: All participants who were randomized and administered at least 1 dose of study drug (Safety Population) and with evaluable basal/parabasal cells data.
  percent of cells
    number analyzed (Participants) | 266 | 262 | 132 | 660
    (all) | 34.4 (35.1) | 31.5 (34.8) | 36.3 (34.3) | 34.1 (34.7)
Percent of Intermediate Cells [Mean (Standard Deviation); unit: percent of cells] — Population: All participants who were randomized and administered at least 1 dose of study drug (Safety Population) and with evaluable intermediate cells data.
  percent of cells
    number analyzed (Participants) | 266 | 262 | 132 | 660
    (all) | 64.7 (34.5) | 67.5 (34.3) | 62.8 (33.9) | 65 (34.2)
Vaginal pH [Mean (Standard Deviation); unit: pH] | 6.2 (0.8) | 6.2 (0.8) | 6.1 (0.7) | 6.2 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Identified as a Responder After Completing Study Treatment in the Generic Estradiol Vaginal Cream and Estrace Vaginal Cream Groups
Description: Treatment comparison of the number of participants in the PP population that were identified as responders at the end of the treatment period evaluated on Day 8 + 1 is presented. A responder was defined as a participant with at least a 25% reduction from baseline in the sum of percent basal/parabasal + percent intermediate cells on vaginal cytology and vaginal pH ≤5.0 with a change from baseline vaginal pH of at least 0.5. Any participant who withdrew from the study because of lack of efficacy was included as a non-responder.
Time Frame: Up to Day 9
Population: Participants who met I/E criteria, didn't develop a concurrent vaginal infection, completed Day 8 visit, and took 6-8 doses and didn't miss >1 dose of study drug (PP Population). As pre-specified in the protocol, only the active groups (Generic Estradiol Vaginal Cream USP, 0.01% and Estrace Vaginal Cream USP, 0.01%) were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Generic Estradiol Vaginal Cream USP, 0.01% | Estrace Vaginal Cream USP, 0.01%
Number analyzed (Participants) | 244 | 227
Participants | 49 | 44
Statistical Analysis 1: Comparison: Generic Estradiol Vaginal Cream USP, 0.01% vs Estrace Vaginal Cream USP, 0.01%; Therapeutic equivalence of the generic estradiol vaginal cream group to the Estrace Vaginal Cream group based on the primary endpoint was evaluated in the PP population; Test type: Equivalence — If the adjusted 90% confidence interval on the difference between proportions of participants considered Responders in the generic estradiol vaginal cream group and the Estrace Vaginal Cream group was contained within the equivalence range [-0.20, +0.20], then treatment with generic estradiol vaginal cream and treatment with Estrace Vaginal Cream were considered therapeutically equivalent; Odds Ratio (OR) = 0.7, 90% CI 2-sided [-5.8 to 7.2]

2. Primary Outcome: Number of Participants Identified as a Responder After Completing Study Treatment in the Generic Estradiol Vaginal Cream, Estrace Vaginal Cream, and Vehicle Vaginal Cream Groups
Description: Treatment comparison of the number of participants in the mITT population that were identified as responders at the end of the treatment period evaluated on Day 8 + 1 is presented. A responder was defined as a participant with at least a 25% reduction from baseline in the sum of percent basal/parabasal + percent intermediate cells on vaginal cytology and vaginal pH ≤5.0 with a change from baseline vaginal pH of at least 0.5.
Time Frame: Up to Day 9
Population: Participants in the PP population, administered at least 1 dose of study drug, and had a post-randomization evaluation (mITT Population). Participants who discontinued early for reasons other than efficacy were included in the mITT population using Last Observation Carried Forward (LOCF).
Measure: Count of Participants; unit: Participants
Arm/Group | Generic Estradiol Vaginal Cream USP, 0.01% | Estrace Vaginal Cream USP, 0.01% | Vehicle Vaginal Cream
Number analyzed (Participants) | 267 | 262 | 132
Participants | 53 | 53 | 0
Statistical Analysis 1: Comparison: Generic Estradiol Vaginal Cream USP, 0.01% vs Vehicle Vaginal Cream; Superiority of the generic estradiol vaginal cream group and the Estrace Vaginal Cream group to the vehicle vaginal cream group based on the primary endpoint was evaluated in the mITT population; Test type: Superiority — The proportion of participants considered as Responders in the generic estradiol vaginal cream group and the Estrace Vaginal Cream group were each compared to the proportion of Responders in the vehicle vaginal cream group. If both the generic estradiol vaginal cream group and the Estrace Vaginal Cream group demonstrated a statistically significant greater proportion of Responders than the vehicle vaginal cream group, then superiority was concluded; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 19.9
Statistical Analysis 2: Comparison: Estrace Vaginal Cream USP, 0.01% vs Vehicle Vaginal Cream; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 20.2

3. Secondary Outcome: Number of Participants Identified as Treatment Success After Completing Study Treatment in the Generic Estradiol Vaginal Cream and Estrace Vaginal Cream Groups
Description: The number of participants in the PP population that are identified as Treatment Success at the end of the treatment period evaluated on Day 8 ± 1 is presented. A Treatment Success is defined as a score of 0 or 1 at Day 8 ± 1 for the symptom identified at baseline as the most bothersome. This evaluation was based on participant self-assessed symptoms of vulvar and vaginal atrophy on a scale of 0 to 3 where 0 = none and 3 = severe. The symptoms that were evaluated were vaginal dryness, vaginal/vulvar irritation/itching, dysuria, vaginal pain associated with sexual activity, and vaginal bleeding. Any participant who withdrew from the study because of lack of efficacy was included as a non-responder.
Time Frame: Up to Day 9
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Generic Estradiol Vaginal Cream USP, 0.01% | Estrace Vaginal Cream USP, 0.01%
Number analyzed (Participants) | 244 | 227
Participants | 161 | 153
Statistical Analysis 1: Comparison: Generic Estradiol Vaginal Cream USP, 0.01% vs Estrace Vaginal Cream USP, 0.01%; Therapeutic equivalence of the generic estradiol vaginal cream group to the Estrace Vaginal Cream group based on the secondary endpoint was evaluated in the PP population; Test type: Equivalence — If the adjusted 90% confidence interval on the difference between proportions of participants considered Treatment Success in the generic estradiol vaginal cream group and the Estrace Vaginal Cream group was contained within the equivalence range [-0.20, +0.20], then treatment with generic estradiol vaginal cream and treatment with Estrace Vaginal Cream were considered therapeutically equivalent; Odds Ratio (OR) = -1.4, 90% CI 2-sided [-9.0 to 6.2]

4. Secondary Outcome: Number of Participants Identified as Treatment Success After Completing Study Treatment in the Generic Estradiol Vaginal Cream, Estrace Vaginal Cream, and Vehicle Vaginal Cream Groups
Description: The number of participants in the mITT Population that are identified as Treatment Success at the end of the treatment period evaluated on Day 8 ± 1 is presented. A Treatment Success is defined as a score of 0 or 1 at Day 8 ± 1 for the symptom identified at baseline as the most bothersome. This evaluation is to be based on participant self-assessed symptoms of vulvar and vaginal atrophy on a scale of 0 to 3 where 0 = none and 3 = severe. The symptoms that were evaluated were vaginal dryness, vaginal/vulvar irritation/itching, dysuria, vaginal pain associated with sexual activity, and vaginal bleeding.
Time Frame: Up to 9 months
Population: Participants in the PP population, administered at least 1 dose of study drug, and had a post-randomization evaluation (mITT Population). Participants who discontinued early for reasons other than efficacy were included in the mITT population using LOCF.
Measure: Count of Participants; unit: Participants
Arm/Group | Generic Estradiol Vaginal Cream USP, 0.01% | Estrace Vaginal Cream USP, 0.01% | Vehicle Vaginal Cream
Number analyzed (Participants) | 267 | 262 | 132
Participants | 175 | 169 | 80
Statistical Analysis 1: Comparison: Generic Estradiol Vaginal Cream USP, 0.01% vs Vehicle Vaginal Cream; Superiority of the generic estradiol vaginal cream group and the Estrace Vaginal Cream group to the vehicle vaginal cream group based on the secondary endpoint was evaluated in the mITT population; Test type: Superiority — The proportion of participants considered as Treatment Success in the generic estradiol vaginal cream group and the Estrace Vaginal Cream group were each compared to the proportion of Treatment Success in the vehicle vaginal cream group. If both the generic estradiol vaginal cream group and the Estrace Vaginal Cream group demonstrated a statistically significant greater proportion of Treatment Success than the vehicle vaginal cream group, then superiority was concluded; p = 0.2897, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 4.9
Statistical Analysis 2: Comparison: Estrace Vaginal Cream USP, 0.01% vs Vehicle Vaginal Cream; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.4949, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 3.9

ADVERSE EVENTS:
Time Frame: Baseline up to Day 9
Description: All participants who were randomized and administered at least 1 dose of study drug (Safety Population).
Arm/Group | Generic Estradiol Vaginal Cream USP, 0.01% | Estrace Vaginal Cream USP, 0.01% | Vehicle Vaginal Cream
All-Cause Mortality (participants affected / at risk) | 0/267 | 0/262 | 0/132
Serious Adverse Events (participants affected / at risk) | 0/267 | 1/262 | 0/132
Other Adverse Events (participants affected / at risk) | 63/267 | 74/262 | 25/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Generic Estradiol Vaginal Cream USP, 0.01% (N=267) | Estrace Vaginal Cream USP, 0.01% (N=262) | Vehicle Vaginal Cream (N=132)
Device occlusion (General disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Generic Estradiol Vaginal Cream USP, 0.01% (N=267) | Estrace Vaginal Cream USP, 0.01% (N=262) | Vehicle Vaginal Cream (N=132)
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1
Retinal tear (Eye disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 0
Application site warmth (General disorders) | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0
Bacterial vaginosis (Infections and infestations) | 2 | 1 | 0
Mucosal excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 1
Adnexa uteri pain (Reproductive system and breast disorders) | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 3 | 8 | 0
Abdominal pain (Gastrointestinal disorders) | 9 | 10 | 3
Abdominal pain lower (Gastrointestinal disorders) | 7 | 3 | 0
Abdominal tenderness (Gastrointestinal disorders) | 4 | 3 | 0
Anorectal discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Cyclic vomiting syndrome (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 1 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Chest discomfort (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 0 | 2 | 0
Discomfort (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 2 | 0
Pain (General disorders) | 1 | 0 | 2
Pyrexia (General disorders) | 1 | 0 | 0
Breast abscess (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 2 | 0
Genital herpes (Infections and infestations) | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1
Otitis media (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 1
Tooth infection (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Carotid bruit (Investigations) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 0
Headache (Nervous system disorders) | 4 | 5 | 2
Migraine (Nervous system disorders) | 0 | 2 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Micturition Urgency (Renal and urinary disorders) | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 0
Breast tenderness (Reproductive system and breast disorders) | 13 | 9 | 1
Endometrial thickening (Reproductive system and breast disorders) | 0 | 1 | 0
Nipple pain (Reproductive system and breast disorders) | 2 | 4 | 0
Pelvic discomfort (Reproductive system and breast disorders) | 1 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 3 | 0
Perineal pain (Reproductive system and breast disorders) | 0 | 1 | 0
Uterine spasm (Reproductive system and breast disorders) | 1 | 2 | 0
Uterine tenderness (Reproductive system and breast disorders) | 0 | 2 | 0
Vaginal erosion (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginismus (Reproductive system and breast disorders) | 1 | 0 | 0
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 1 | 3 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 | 4 | 1
Vulvovaginal erythema (Reproductive system and breast disorders) | 1 | 0 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 1 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 2 | 2 | 1
Vulvovaginal swelling (Reproductive system and breast disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pterygium operation (Surgical and medical procedures) | 0 | 0 | 1
Sinus operation (Surgical and medical procedures) | 0 | 1 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 0 | 0
Flushing (Vascular disorders) | 1 | 1 | 0
Hot flush (Vascular disorders) | 1 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed.

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-08-04): https://cdn.clinicaltrials.gov/large-docs/38/NCT03294538/SAP_000.pdf
  • Study Protocol (2016-04-18): https://cdn.clinicaltrials.gov/large-docs/38/NCT03294538/Prot_001.pdf